CLINICAL TRIAL: NCT03284060
Title: Social Cognition Training and Cognitive Remediation : a New Tool for 22q11.2 Deletion Syndrome
Brief Title: Social Cognition Training and Cognitive Remediation
Acronym: RCKID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulties
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A00881-52
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: 22q11.2 Deletion Syndrome
Keywords: Cognitive remediation, 22q11.2 deletion syndrome
MeSH Terms: conditions — DiGeorge Syndrome

STUDY DESIGN:
Intervention Model Description: open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive remediation program (Experimental)
  Interventions: Behavioral: Cognitive remediation program

INTERVENTIONS:
Behavioral: Cognitive remediation program — Cognitive remediation program is a set of reeducation techniques and aims at restoring or compensating altered cognitive functions such as memory, attentional or executive functions, and social cognition. Therapists help individuals develop new information processing strategies designed to meet their needs and wishes. Specific therapeutic sessions are designed to generalize such strategies to everyday situations to reduce the impact of cognitive deficits on daily life. Thus, social cognitive training therapy helps the development of personal strategies specifically adapted to preserve skills and reduce the difficulties.
  16 sessions (45 min) of cognitive remediation with the therapist are proposed, each session is composed of three parts:
  1. pen and paper tasks focusing on specific emotion recognition component (20 min),
  2. computerized tasks focusing on the same process (20 min),
  3. a proposal of a home-based task (during 20 min).

SUMMARY:
Social cognition refers to mental operations that enable people to perceive, interpret constantly changing social informations. These processes allow people to rapidly, effortlessly and flexibly perceive and interpret rapidly-changing social information, and respond appropriately to social stimuli. Besides, this ability gives meaning to the actions of others. Impairments in this field may largely underlie social dysfunctions and reduce adaptive skills. Moreover, social cognitive disabilities contribute more or less directly to behavioral disturbances and psychiatric symptoms The "RC KID" program involves a variety of exercises in a paper and/or pencil or a computerized format or role playing and a strategy coaching approach. "RC KID" targets the emotion recognition and social interaction.

A little cartoon character (a pirate), is supposed to be very friendly and kind toward children. The pirate will accompany them throughout the program for an effective and positive reinforcement. The main goal of "RC KID" is to adjust to children's difficulties in daily life.

Moreover, since the cognitive remediation benefit is complex to apply in daily life, the program is based on a metacognitive strategy.

After a complete neuropsychological assessment and a psychoeducational session (with the child and the parents), 16 1-h-sessions of cognitive remediation with the therapist are proposed. Each session is composed of three parts: (1) computerized tasks focusing on specific emotion recognition components (20 min). RC KID is composed of 2 modules : Emotion recognition and social interaction. These tasks contain photo or video. (2) pen and paper or role playing tasks focusing on the same processes (20 min) (3) a proposal of a home-based task (during 20 min). Weekly, home tasks are proposed to the child and analyzed with the parents and the therapist. Indeed, home exercises are useful to promote the transfer of strategies to daily life and their subsequent automation. The heterogeneity of cognitive deficits in 22q11.2 deletion necessitates an individualized cognitive remediation therapy. In this regard, "RC KID" seems to be a promising tool.

DETAILED DESCRIPTION:
The second objective is to evaluate the impact of RC KID on behavior disorders. Method : a validation study using multiple single-case experimental designs. A thorough assessment, including a complete evaluation of components of social cognition but also clinical and neuropsychological assessments is proposed for each patient enrolled in the study.

Investigators collect three kinds of baselines before the beginning of the cognitive remediation intervention: baselines specific of the targeted component (Emotion recognition and Theory of Mind), non-specific baselines (such as measures of neurocognition processes that should not be affected by the intervention), and intermediary baselines that is measures of social cognitive function linked with targeted processes but not directly concerned by the cognitive remediation program.

These measures and the complete assessment will be repeated at the end of the intervention to highlight impacts of RC KID on social cognitive impairments, and 6 months later to investigate the possible long-lasting effects of the benefits.

ELIGIBILITY:
Inclusion Criteria:

* Children with diagnosis of 22q11.2 deletion syndrome (CGH-Array and FISH)
* Native French speaker
* Clinically stable
* Parental and children consent

Exclusion Criteria:

* history of neurological illness or trauma
* Taking of medicine with somatic aim having a cerebral or psychic impact
* Simultaneous participation on another program of cognitive remediation
* child or parents unlikely to cooperate

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the variation in sub-scores of specific baselines, obtained before and after cognitive remediation intervention: | 6 months
  baselines specific of the targeted component (Emotion recognition and Theory of Mind), non-specific baselines (such as measures of neurocognition processes that should not be affected by the intervention), intermediary baselines that is measures of social cognitive function linked with targeted processes but not directly concerned by the cognitive remediation program.
  These measure is repeated at the end of the intervention to highlight the impact of the " RCKID " program, and 6 months later to investigate the possible long-lasting effects of the benefits

SECONDARY OUTCOMES:
Aberrant Behavior Checklist scale | 6 months
  Change in sub-score " hyperactivity / non compliance " (scale " Aberrant Behavior Checklist ") (completed by parents or the educational team). This measure is repeated at the end of the intervention to highlight the impact of the " RC KID " program, and 6 months later to investigate the possible long-lasting effects of the benefits.
MDI-C scale ( Multiscore Depression Inventory for Children scale) | 6 months
KIDSCREEN-27 scale | 6 months
  The KIDSCREEN-27 with five dimensions resulted. All five dimensions are Rasch scales: Physical Well-Being (5 items), Psychological Well-Being (7 items), Autonomy & Parents (7 items), Peers & Social Support (4 items), and School Environment (4 items).
Vineland 2 scale (Vineland Adaptive Behavior Scale) | 6 months
  A measure of adaptive behavior from birth to adulthood

CONTACTS AND LOCATIONS:
Overall Officials: DEMILY CAROLINE, PH, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Hopital Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No